CLINICAL TRIAL: NCT04358913
Title: Northern Alberta Linac-MR Image-Guided Human Clinical Trials - 1
Brief Title: MR Imaging Study Using the Northern Alberta Linac-MR (Northern LIGHTs - 1)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IIT-0013
Record Dates: First submitted 2020-04-09; First posted 2020-04-24 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MR Imaging on the Alberta linac-MR P3 system (Experimental): All participants will undergo a single MR imaging session (30-40 minutes) on the Alberta linac-MR P3 system.
  Interventions: Device: MR scan with the Alberta linac-MR P3 system

INTERVENTIONS:
Device: MR scan with the Alberta linac-MR P3 system — Single MR imaging session to develop and optimize the necessary MR sequences on the Alberta linac-MR P3 system to allow for MR-guided radiotherapy.

SUMMARY:
Cancers are often treated with external beam radiotherapy. Current radiotherapy treatments are performed using computed tomography (also known as CT) scans which may not always clearly identify the cancer. In some instances, magnetic resonance imaging (MRI) may be able to better identify cancers. Therefore, efforts are currently underway to use the MRI scans to improve radiotherapy treatments or eventually even use radiotherapy equipment that only uses MRI scans to guide treatments. This new technology that will only use MRI scans to guide treatments is called the Linac-MR (linear accelerator with an MRI). The purpose of this pilot phase of the study is to test whether the Alberta linac-MR P3 system at the Cross Cancer Institute can acquire high quality MR images safely. It will allow the researchers to develop the best collection of MR images possible with this new machine, in order to allow them to visualize tumors for future patients that are treated on this machine.

DETAILED DESCRIPTION:
This prospective, pilot phase, clinical trial is an imaging study to optimize the necessary MR sequences on the Alberta linac-MR P3 system to allow for MR-guided radiotherapy in adult patients with cancer that are treated with high dose external beam radiotherapy. Each participant will undergo a single MR imaging session (30 - 40 minutes) on the Alberta linac-MR P3 system. Towards the end of the study, patients will be approached to participate in an optional sub-study, where they will undergo a total of five MR imaging sessions (performed every two to five days) to allow for an assessment of inter-fraction motion.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Patients deemed fit to undergo high dose external beam radiation therapy by their attending radiation oncologist

Exclusion Criteria:

* Patients with contraindications for MRI
* Patients who are unable to lie flat and still for the duration of the expected scan acquisition
* Patients who are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Number of high-quality MR image data sets acquired for each major tumour site (prostate, liver, lung, CNS, breast, gynecological, pancreas, and head and neck) | Through study completion, approximately 7 years
  Clinical radiologists, medical physicists, and radiation oncologists will work together to develop MR sequences that can delineate tumour target volumes on the Alberta linac-MR P3 system. Over the course of the trial, the clinical radiologists will work with medical physicists to optimize these sequences to allow for the development of optimal MR images, with the goal to develop of series of protocols that can be utilized to provide clear MR image guidance for each tumour group.

SECONDARY OUTCOMES:
Quantify the patient experience on the Linac-MR | After the first and last scan, up to 5 weeks
  Participants will complete a questionnaire at the end of their first scan regarding their experience having imaging done on the Linac-MR. Participants taking part in the optional sub-study will complete the same questionnaire at the end of their last set of imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Nawaid Usmani, MD, Principal Investigator — Cross Cancer Institute, Alberta Health Services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No